CLINICAL TRIAL: NCT07340879
Title: Reconstruction of Orbital Floor Blow-out Fractures by Titanium Mesh Versus Autogenous Iliac Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Menatallah Gamal Saleh, lecturer of ophthalmology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-2023-300338
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Blow-Out Fractures
Keywords: Orbital fractures; titanium mesh; blow-out
MeSH Terms: conditions — Orbital Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with orbital blow-out fractures (Active Comparator): Treated by immediate surgical reconstruction of orbital floor blow-out fractures by titanium mesh (within 2 week of the trauma)
  Interventions: Procedure: Titanium mesh
- Patients with orbital blow-out fractures were selected irrespective of their age and gender (Active Comparator): Treated by immediate reconstruction of orbital floor by autogenous iliac graft (within 2 week of the trauma)
  Interventions: Procedure: autogenous iliac graft

INTERVENTIONS:
Procedure: Titanium mesh — Insertion of prefabricated titanium mesh to close the defect in the orbital floor
  Arms: Patients with orbital blow-out fractures
Procedure: autogenous iliac graft — Incision over the iliac bone to take iliac bone graft which cover the defect in the orbital floor that is measured intraoperatively.
  Arms: Patients with orbital blow-out fractures were selected irrespective of their age and gender

SUMMARY:
Blow-out fractures result from direct blunt impacts to the orbit which causes an immediate rise increase in intra-orbital pressure. Decompression via fracture of the orbital floor then occurs. Motor vehicle accidents are the main cause of orbital trauma. Also, industrial accidents, sports-related facial trauma, and assaults are important causes.

Clinical manifestations include ecchymosis, limitation of eye movements resulting in diplopia, enophthalmos. Very rarely, severe pain and nausea immediately after the injury are reported.

Radiologic evaluation including computed tomography (CT), plane radiology and magnetic resonance imaging (MRI) are the mainstay diagnostic modalities used for evaluation of cases with orbital trauma.

Treatment of the orbital blow-out fractures is aimed at restoring floor continuity, thus providing adequate support for orbital contents preventing their herniation and incarceration, thereby possible subsequent fibrosis of soft tissues most importantly extraocular muscles.

Various alloplastic or autogenous grafts are used for reconstruction of orbital blow-out fractures.

DETAILED DESCRIPTION:
A prospective interventional randomized controlled study, including 80 patients (who presented at trauma unit in Assiut university hospital between May 2020 to May 2023 and fulfilled the inclusion criteria) was conducted. Patients with orbital floor blow-out fractures were selected irrespective of their age and gender. The study followed the tenets of the Helsinki declaration and guidelines of the local research committee. An informed written consent was signed by all the patients who agreed to be enrolled in the study, or their relatives if consciously disturbed patients. All operations were done within 2 weeks of the trauma.

Patients were divided into 2 groups:

* Group I (40 patients) consists of immediate surgical reconstruction of pure orbital floor blow-out fractures by titanium mesh.
* Group II (40 patients) consists of immediate surgical reconstruction of pure orbital floor blow-out fractures by autogenous iliac graft.

Inclusion criteria:

Clinical Enophthalmos, diplopia, and/or limited ocular motility in one or more directions.

Radiological:

- CT scan (axial, coronal & 3 dimensional):

Fracture of the orbital floor with herniation of the orbital contents (extra-ocular muscles, or orbital fat).Exclusion criteria:

patients with bilateral orbital fractures or severe facial fractures. Also, patients with bad general condition or uncontrolled diabetes mellitus were excluded.

Ophthalmological examination of study subjects was performed by an expert ophthalmologist (MGA). This included examination of the anterior segment and evaluation of pupillary reflexes by penlight and slit lamp to document associated eye globe injuries. Fundus examination was carried out using binocular indirect ophthalmoscope. Also, measurement of the corrected distance visual acuity (CDVA) expressed as decimal notation using a chart projector utilizing built in Snellen's charts. Also, ocular motility examination in the six cardinal positions of eye movements was carried out to document any limitation of eye movement (direction and degree). Moreover, Hertel's exophthalmometer was used to measure the degree of enophthalmos in the involved eye. A difference of 2 or more millimeters between both eyes was considered significant for enophthalmos in the sunken eye. Ophthalmological features of study subjects. Postoperative care

* A head-up position was adopted by patients in the early postoperative period with application of cold compresses in order to reduce postoperative edema.
* Analgesia and antibiotics were prescribed.

Follow up:

Follow-up examinations to assess visual acuity, extra-ocular motility, pupillary reaction. Also, the degree of enophthalmos was measured. Assessment of sensation over the check to assess the degree of neuralgia and patients were asked about improvement in double vision. Those parameters were monitored for at least 6 months after surgery and up to one year.

Follow up orbital CT scan (coronal view was done for all patients in the study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Enophthalmos, diplopia, and/or limited ocular motility in one or more directions.

Radiological:

- CT scan (axial, coronal & 3 dimensional): Fracture of the orbital floor with herniation of the orbital contents (extra-ocular muscles, or orbital fat)

Exclusion Criteria:

* patients with bilateral orbital fractures or severe facial fractures.
* Patients with bad general condition or uncontrolled diabetes mellitus.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-05-02 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Assess visual acuity, extra-ocular motility, pupillary reaction. Also, the degree of enophthalmos | 1 year
  CDVA expressed as decimal notation using a chart projector utilizing built in Snellen's charts. Also, ocular motility examination in the six cardinal positions of eye movements was carried out to document any limitation of eye movement (direction and degree). Moreover, Hertel's exophthalmometer was used to measure the degree of enophthalmos.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Assiut, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim YS, Kim JH, Hwang K. The Frequency of Decreased Visual Acuity in Orbital Fractures. J Craniofac Surg. 2015 Jul;26(5):1581-3. doi: 10.1097/SCS.0000000000001860. PMID 26114513
- [Background] Jordan DR, Allen LH, White J, Harvey J, Pashby R, Esmaeli B. Intervention within days for some orbital floor fractures: the white-eyed blowout. Ophthalmic Plast Reconstr Surg. 1998 Nov;14(6):379-90. doi: 10.1097/00002341-199811000-00001. PMID 9842557
- [Background] Bord SP, Linden J. Trauma to the globe and orbit. Emerg Med Clin North Am. 2008 Feb;26(1):97-123, vi-vii. doi: 10.1016/j.emc.2007.11.006. PMID 18249259